CLINICAL TRIAL: NCT04329598
Title: The Effects of Whole-Body Electromyostimulation Application on Balance, Pain, Physical Conformity Parameters and Quality of Life in Individuals With Lumbar Disc Hernia: a Comperative Study
Brief Title: Effects of Whole-Body Electromyostimulation Application in Individuals With Lumbar Disc Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Alp Eşrefoğlu, Physiotherapist, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/23-07
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Lumbar Disc Herniation
Keywords: Whole body electromyostimulation; Lumbar disc herniation; Balance; Pain; Physical Conformity Parameters; Quality of Life
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain

STUDY DESIGN:
Intervention Model Description: A Comparative Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-Body Electromyostimulation Group (Experimental): Whole-Body Electromyostimulation group includes exercises with electric stimulation. Whole-Body Electromyostimulation group will have 45 minutes of exercises which are specific exercises for Lumbar Disc Herniation.
  Interventions: Other: Whole-Body Electromyostimulation Group
- Exercise Group (Experimental): Exercise group includes exercises without electric stimulation. Exercise group will have 45 minutes of exercises which are specific exercises for Lumbar Disc Herniation.
  Interventions: Other: Exercise Group

INTERVENTIONS:
Other: Whole-Body Electromyostimulation Group — Whole-Body Electromyostimulation group includes exercises with electric stimulation. Whole-Body Electromyostimulation group will have 45 minutes of exercises which are specific exercises for Lumbar Disc Herniation.
  Arms: Whole-Body Electromyostimulation Group
Other: Exercise Group — Exercise group includes exercises without electric stimulation. Exercise group will have 45 minutes of exercises which are specific exercises for Lumbar Disc Herniation.
  Arms: Exercise Group

SUMMARY:
To determine the effects of WB-EMS application on balance, pain, muscle strength, muscle endurance, flexibility, muscle shortening and quality of life in individuals with Lumbar Disc Hernia and compare it with individuals who have not received this training.

DETAILED DESCRIPTION:
Lumbar disc hernia (LDH); It is one of the common spinal problems that occur in the form of low back pain and radiculopathy that spreads to the lower extremities. The prevalence of lumbar disc herniation reported in individuals with low back pain; It ranges from 0% to 47%. It has been reported that the highest prevalence of LDH is in adults between the ages of 30-50. Disc herniation at the L4-5 and L5 - S1 spinal levels is more common in adults over the age of 55. The most important complaint in LDH is pain, and patients often complain of a blunt pain in the lumbar region. Weakness in the muscles surrounding the vertebra can cause balance and walking problems. For Lumbar Disc Hernia, sedentary life, gender, high body mass index, occupation, smoking, psychosocial factors and people exposed to vibration for a long time are among the risk factors. Lack of time is reported to be the biggest obstacle to exercising. In addition, kinesiophobia, that is the fear of pain due to movement, is very common in this group. Physical activity and exercise are arguably the most comprehensive therapeutic agent for a long-term and fundamentally established society. There is a consensus on the review of the current literature that it positively affects the risk of exercise disease, but not all, risk factors, diseases, and disability between middle and advanced age. Whole Body Electromyostimulation (WB-EMS), a technology that addresses nine (main) muscle groups, may be a good option. Given the low training intensity of 1-2 sessions per week for 20 sessions, it may be of interest to people who are close to traditional exercise programs, with low volunteer intensity and a high degree of oversight and individualization of existing WB-EMS settings.

ELIGIBILITY:
Inclusion Criteria:

* Bulging or protruding disc herniation between L1-S1 levels diagnosed by the attending physician
* Without a neurological sign
* Not attending physiotherapy and rehabilitation session in the last 6 months
* No regular exercise habits
* No previous WB-EMS experience

Exclusion Criteria:

* Use of muscle relaxants
* Pain medication use
* Pacemaker
* Implants
* Having a history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Y Balance test | 8 weeks
  The assessor should place his fingers behind the line to stand on the platform and should be instructed to push the access indicator in the target area in the tested direction. After three attempts with each member in each direction, the evaluator checks whether the individual has performed at least one successful test. Otherwise, the evaluator will request an additional test until the interval is correct. This test is evaluating dinamic balance.
Static balance evaluation | 8 weeks
  Both feet will be recorded for one-foot standing times for static balance assessment. Individuals will be asked to stand in one-foot standing position with their hands at the waist and stand for as long as they can. Each evaluation will be done in 3 replications and the best result will be recorded.

SECONDARY OUTCOMES:
Oswestry Disability Index | 8 weeks
  Oswestry Disability Index (ODi) was used to determine the degree of disability. ODI consists of 10 items that measure the severity of pain, personal care, lifting, walking, sitting, standing, social life, sleep and pain. Each item is rated between 0-5. As the total score increases, the level of disability increases. The maximum score is 50 points; 31-50 points are considered heavy, 11-30 points are moderate and 1-10 points are considered light. By converting the total score obtained from the patient to the percentile system, the percentage of disability will be calculated.
Pain assessment | 8 weeks
  First Part: In this section, the patient is asked to mark the location of the pain on the body diagram and indicate "D" if the pain is coming deeply, "Y" on the body surface and "DY" on both the deep and the surface. Second Part: In this part, there are 20 sets of word groups that examine pain in terms of sensory, perceptual and evaluation. Each group consists of 2-6 words that describe pain with different aspects. The patient is told to select the word set that matches his pain and mark the word that matches his pain in the chosen set. The first 10 of the 20 word sets in the second part of the MASF include the sensory size of the pain, the next five clusters perceptual dimension, and the 16th set includes the assessment. The last four clusters are composed of words that show various aspects of pain. Part Three: This section includes the relationship of pain over time. There are groups of words to determine the continuity, frequency, and factors that increase / decrease pain.
Muscle strengtening test | 8 weeks
  Hand Held Dynamometer is used to measure isometric muscle strength of upper limb, lower limb and trunk muscles. This measurement is repeated 2 times for each muscle and the average of the force at the time of their position deterioration is recorded in kilograms. This measurement was repeated 2 times for each direction and the average of the force at the moment the position was broken will be recorded in kilograms.
Muscle endurance test | 8 weeks
  This test is performed to evaluate the endurance of the muscle group evaluated. After giving the appropriate position to the muscle group to be evaluated, the person is asked to protect as much as he can maintain that position and it is recorded in seconds.
Muscle shortness test | 8 weeks
  With this test, muscle shortness will be evaluated. After giving the appropriate position to individuals, measurements will be taken using goniometer and tape measure and the data will be recorded. These muscles are pectoral muscle, hamstrings, hip flexor muscles, quadriceps and lumbar extensor muscles
Evaluation of flexibility | 8 weeks
  Sit and reach test: The patients were asked to take a long sitting position on the floor. Metric scale placed on the tip of the soles of the foot in this position they were asked to reach forward on the scale found of cases the longest distance they can reach is noted in centimeters Trunk lateral flexion test: In measurement, feet are adjacent, arms are freely trunk measurement was made next to it. First, the outer surface of the thigh of the distal end of the right hand the place on it was determined, then sliding his hands down from the dancers they were asked to bend their body sideways. With the maximum point that cases can go The difference between the resting position is noted in centimeters. Measurement left repeated for the side
Assessment of quality of life | 8 weeks
  Short Form-36 (SF-36) is a self-assessment scale and 36 items of 8 dimensions of health such as physical function, social function, role restrictions (due to physical and emotional causes), mental health, vitality (energy), pain and general perception of health.

CONTACTS AND LOCATIONS:
Overall Officials: Alp Esrefoglu, PT, Principal Investigator — Eastern Mediterranean University; Ender Angın, PhD, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean Üniversity, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kemmler W, Weissenfels A, Willert S, Shojaa M, von Stengel S, Filipovic A, Kleinoder H, Berger J, Frohlich M. Efficacy and Safety of Low Frequency Whole-Body Electromyostimulation (WB-EMS) to Improve Health-Related Outcomes in Non-athletic Adults. A Systematic Review. Front Physiol. 2018 May 23;9:573. doi: 10.3389/fphys.2018.00573. eCollection 2018. PMID 29875684
- [Background] Kemmler W, Weissenfels A, Bebenek M, Frohlich M, Kleinoder H, Kohl M, von Stengel S. Effects of Whole-Body Electromyostimulation on Low Back Pain in People with Chronic Unspecific Dorsal Pain: A Meta-Analysis of Individual Patient Data from Randomized Controlled WB-EMS Trials. Evid Based Complement Alternat Med. 2017;2017:8480429. doi: 10.1155/2017/8480429. Epub 2017 Oct 18. PMID 29234437
- [Background] Weissenfels A, Teschler M, Willert S, Hettchen M, Frohlich M, Kleinoder H, Kohl M, von Stengel S, Kemmler W. Effects of whole-body electromyostimulation on chronic nonspecific low back pain in adults: a randomized controlled study. J Pain Res. 2018 Sep 20;11:1949-1957. doi: 10.2147/JPR.S164904. eCollection 2018. PMID 30288089